CLINICAL TRIAL: NCT05832697
Title: An Exploratory Clinical Trial to Evaluate and Compare Safety and Pharmacokinetic Characteristics After Administration of the DWJ1439, DWJ1464, DWC202108 or DWC202109 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1464103
Record Dates: First submitted 2023-04-02; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Ursodeoxycholic Acid; Tablets

STUDY DESIGN:
Intervention Model Description: 4 by 3 cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Active Comparator): P1: DWJ1439(ursodeoxycholic acid) 100mg, P2: DWC202108(usrodeoxycholic acid) 250mg, P3: DWJ1464(ursodeoxycholic acid) 100mg
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Tablet
- Treatment B (Active Comparator): P1: DWC202108(usrodeoxycholic acid) 250mg, P2: DWJ1439(ursodeoxycholic acid) 100mg, P3: DWC202109(ursodeoxycholic acid) 250mg
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Tablet
- Treatment C (Active Comparator): P1: DWJ1464(ursodeoxycholic acid) 100mg, P2: DWC202109(ursodeoxycholic acid) 250mg, P3: DWJ1439(ursodeoxycholic acid) 100mg
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Tablet
- Treatment D (Active Comparator): P1: DWC202109(ursodeoxycholic acid) 250mg, P2: DWJ1464(ursodeoxycholic acid) 100mg, P3: DWC202108(usrodeoxycholic acid) 250mg
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Tablet

INTERVENTIONS:
Drug: Ursodeoxycholic Acid 250 Mg Oral Tablet — Administration of Ursodeoxycholic Acid 250 Mg Oral Tablet or Ursodeoxycholic Acid 100 Mg Oral Tablet
  Other Names: Ursodeoxycholic Acid 100 Mg Oral Tablet

SUMMARY:
This study aims to Evaluate and Compare Safety and Pharmacokinetic Characteristics after Administration of the DWJ1439, DWJ1464, DWC202108 or DWC202109 in Healthy Adult Volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to explore the differences in pharmacokinetics and safety characteristics between Test Drugs(DWJ1439, DWJ1464) and that of Reference Drugs(DWC202108, DWC202109) in healthy adults with fasting state: Randomized, open-label, oral, single-dose, four-treatment, three-period, non-replicated crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 years old to under 55.
* BMI 18.0≥ and ≤30 kg/m² with body mass ≥50 kg
* Those who have no congenital or chronic disease requiring treatment and have no pathological symptoms or findings as a result of medical examination.
* Those who have no clinically significant abnormalities in general physical examination, laboratory assessments and 12-lead electrocardiogram (ECG).
* Those who understand the requirements of the study and sign a written informed consent, and also accept all the restrictions imposed during the course of the study.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition. Participation in a clinical drug study or bioequivalence study 6 months prior to the present study.
* Refusal to abstain from smoking or consumption of tobacco products 72 hours before drug administration and during each study period.
* Refusal to abstain from caffeine or grapefruit containing food or drinks for 72 hours before drug administration and during each study period.
* Refusal to abstain from strenuous activities for 72 hours before drug administration and post-study visit, before and during each study period.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Baseline corrected/uncorrected ursodeoxycholic acid AUC0-t | -48 - 72hours
  Baseline corrected/uncorrected ursodeoxycholic acid의 AUC0-t
Baseline corrected/uncorrected ursodeoxycholic acid의 Cmax | -48 - 72hours
  Baseline corrected/uncorrected ursodeoxycholic acid의 Cmax
Baseline corrected/uncorrected total ursodeoxycholic acid의 AUC0-t | -48 - 72hours
  Baseline corrected/uncorrected total ursodeoxycholic acid의 AUC0-t
Baseline corrected/uncorrected total ursodeoxycholic acid의 Cmax | -48 - 72hours
  Baseline corrected/uncorrected total ursodeoxycholic acid의 Cmax

CONTACTS AND LOCATIONS:
Overall Officials: BoHyung Kim<bhkim98@gmail.com> Kim, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Medical Hospital, Seoul, Korea, Republic of, South Korea

IPD SHARING:
Plan to Share IPD: Undecided